CLINICAL TRIAL: NCT04559373
Title: A Virtual Reality and Field Training Toolkit to Enhance Community Ambulation and Participation in Stroke Survivors
Brief Title: Virtual Reality and Field Training to Enhance Community Walking After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Jewish Rehabilitation Hospital (Other); Integrated University Health and Social Services Center of the Capitale-Nationale (Other); Laval University (Other)
Responsible Party: Principal Investigator, Anouk Lamontagne, Associate Professor, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PJT-148917
Record Dates: First submitted 2020-07-06; First posted 2020-09-22 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-11

CONDITIONS: Stroke
Keywords: Aging; Biomechanics; Community ambulation; Intervention; Locomotion; Rehabilitation; Sensorimotor integration; Virtual reality
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Intervention study involving a single group, multiple-pre, multiple-post, sequential design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual Reality and Field Practice Training (VRFT) (Experimental): Participants will engage in a 4-week VRFT intervention that comprises of 1-hour training sessions, 3 times/week.
  Interventions: Other: Virtual Reality and Field Training (VRFT)

INTERVENTIONS:
Other: Virtual Reality and Field Training (VRFT) — The VRFT intervention involves the intensive practice of community ambulation skills. Some of the training sessions will be performed in a virtual environment, while others will consist of field training exercises in the community. During the intervention, stroke participants will be invited to practice different dimensions of community ambulation, such as postural transitions, avoiding other pedestrians, dual-task walking, etc.

SUMMARY:
While stroke survivors discharged from rehabilitation present with some recovery in mobility, their ability to ambulate in the community remains limited. The investigators propose to test a novel, low-cost, intensive and individually tailored intervention that combines virtual reality (VR) and field training to enhance community ambulation and participation in stroke survivors discharged from rehabilitation.

The aims are to: (1) Assess feasibility, acceptability, safety and adherence of the intervention in stroke survivors; and (2) Examine the extent to which post-intervention changes in functional walking and participation to community walking vary according to walking, cognitive and visual-perceptual abilities.

The investigators will use a virtual environment prototype simulating a shopping mall and surrounding streets, in which participants will interact using VR goggles and game controllers. Scenarios of increasing levels of complexity will be introduced. This intervention study involves a single group, multiple pre- multiple post- study design where chronic stroke participants will engage in a 4-week training program. The program will include VR training sessions performed in the clinical setting (3/week) and practice of community ambulation skills while supervised by family/caregivers (2/week). Participants will be assessed on measures of functional walking, balance & mobility and participation to community walking. Adherence, safety and acceptability will be documented. This study will generate foundation knowledge on the response to the intervention based on individual capacities.

DETAILED DESCRIPTION:
Ambulating in community environments requires the skills to cope with multiple, simultaneous dimensions such as walking speed and distance, etc. Such skills remain compromised in the majority of stroke survivors due to insufficient or lack of targeted practice. The investigators propose to test a new, individually-tailored intervention, developed by the research team, grounded in best evidence in community ambulation, principles of motor learning and participatory action research. This unique intervention will combine virtual reality (VR) and field training practice to optimize learning that can be generalized to daily walking activities.

Participants will engage in the 4-week, individually-tailored intervention that comprises of supervised VR training sessions (3 times/week) performed in the clinical setting. VR sessions will be completed by field training assignments. Subjects will be assessed twice prior to the intervention, immediately after the intervention and at follow up.

Generalized estimating equations will be used to compare changes in main and secondary outcomes across time points, with each personal factor of interest (e.g. walking capacity, visual-perceptual function, and cognitive function) analyzed individually while adjusting for age. Outcomes on adherence, safety and acceptability will be analyzed with descriptive statistics.

Required sample size was estimated based on Green's rule (effect size=0.5, power=80%, α=0.05) with a variance inflation factor assuming moderate within-subject correlations for 3 post-baseline measurement time points. This yields a sample size of 30. Assuming a worst-case scenario of 30% attrition rate, a total of 40 stroke subjects (20/site) will be recruited.

ELIGIBILITY:
Inclusion Criteria:

People with chronic stroke and persistent deficits in walking / visual-perceptual / cognitive capacities. They can be male or female, aged from 40 to 74 years, with normal/corrected visual and auditory acuity, and present with:

* First-ever supratentorial unilateral stroke 9-24 months ago (such chronicity will ensure steady-state mobility without long-term disuse-related changes
* Mild-to-moderate hemiparesis (Chedoke McMaster Stoke Assessment stages 4/7-6/7 on postural control, leg & foot)
* Ability to walk independently with/without walking aids for at least 1 min at 0.4-0.9 m/s (such a speed range indicates mobility not sufficient for functional community ambulation: shopping ~1.1m/s, street crossing ~1.2 m/s)
* Intact or mildly affected cognitive function (Montreal Cognitive Assessment scores ≥ 22/30)
* Intact to moderately affected visual-perceptual function (positive scores on a maximum of 3/6 tasks on the Behavioural Inattention Test)

Exclusion Criteria:

* Subjects with comorbidities interfering with walking
* Subjects with comorbidities interfering with visual perception
* Subjects without medical clearance for exercise

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-intervention change in the Six Minute Walk Test (6MWT) | Pre-intervention (Week4) and post-intervention (Week8)
  The six-minute walk test measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
Change in the Six Minute Walk Test (6MWT) at Follow-up | Post-intervention (Week8) and Follow-up (Week12)
  The six-minute walk test measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.

SECONDARY OUTCOMES:
Dynamic Gait Index | Baseline (Week0), pre-intervention (Week4), post-intervention (Week8) and follow-up (Week12)
  Developed to assess the likelihood of falling in older adults
5m Walk Test | Baseline (Week0), pre-intervention (Week4), post-intervention (Week8) and follow-up (Week12)
  Assesses walking speed in meters per seconds over a short duration
Activities-Specific Balance Confidence Scale | Baseline (Week0), pre-intervention (Week4), post-intervention (Week8) and follow-up (Week12)
  16-item self-reported measure of balance confidence performing various activities without losing balance or experiencing a sense of unsteadiness. Items are rated on a 0%-100% response scale, with a score of 0 representing no confidence and a score of 100 representing complete confidence.
Trip Activity Log | Baseline (Week0), pre-intervention (Week4), post-intervention (Week8) and follow-up (Week12)
  Questionnaire to record the number of trips and walking-related activities in the community (e.g. outside home) 3 days preceding its administration
Environmental Analysis of Mobility Questionnaire | Baseline (Week0), pre-intervention (Week4), post-intervention (Week8) and follow-up (Week12)
  Self-reported tool to assess mobility problems due to the environment
Assessment of Life Habits (Life-H: mobility and community life domains) | Baseline (Week0), pre-intervention (Week4), post-intervention (Week8) and follow-up (Week12)
  Assesses mobility and community life habits based on the levels of accomplishment and assistance required as well as satisfaction

OTHER OUTCOMES:
Adherence to intervention | 3x/week over the 4-week intervention for the virtual reality component; 2x/week over the 4-week intervention for the field training component
  Training logbook filled by researchers/clinicians (virtual reality) and subjects (field training) component)
Safety of the intervention | 3x/week over the 4-week intervention of the virtual reality component
  Assesses by systematically collecting any occurrence of adverse/unwanted events (falls, injuries, fatigue, etc).
Acceptability of the intervention | Post-intervention (Week8)
  Assesses using the Technology Acceptance Model based Questionnaire (Tam-Q) based on the technology acceptance model, in which subjects will rate their perception on each dimension using a visual analog scale ranging from 0-56, with higher score representing higher acceptance to the intervention.
Cadence | Pre-intervention (Week4) and post-intervention (Week8)
  Cadence is the rate at which a person walks (steps per minute) and will be measured with the GaitRite system.
Step length | Pre-intervention (Week4) and post-intervention (Week8)
  Step length is the distance (in meters) from a point of contact with the ground of one foot to the following occurrence of the same point of contact with the other foot and will be measured with the GaitRite system.
Step duration | Pre-intervention (Week4) and post-intervention (Week8)
  Step duration is the period of time (in seconds) taken for one step is measured from an event of one foot to the following occurrence of the same event with the other foot and will be measured with the GaitRite system.
Stance phase | Pre-intervention (Week4) and post-intervention (Week8)
  Stance phase is the period of time when the foot is in contact with the ground (%) and will be measured with the GaitRite system.
Swing phase | Pre-intervention (Week4) and post-intervention (Week8)
  Swing phase is the period of time when the foot is not in contact with the ground (%) and will be measured with the GaitRite system.

CONTACTS AND LOCATIONS:
Overall Officials: Anouk Lamontagne, PhD, Principal Investigator — McGill University
Locations (2):
- Canada (2):
  - Jewish Rehabilitation Hospital, Laval, Quebec
  - Institut de réadaptation en déficience physique de Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measure will be made available.
Time Frame: Data will be available within 6 months of study completion
Access Criteria: De-identified data will be deposited in a REDCap database and made available to collaborators. Data may also be made available to other researchers via an institutional data repository that will allow adhering to FAIR principles.